CLINICAL TRIAL: NCT05396274
Title: Investigation of the Clinical Efficacy of High Flow Nasal Oxygen in Patients Over 60 Years of Age Undergoing Colonoscopy
Brief Title: High Flow Nasal Oxygen Therapy Undergoing Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Turkish Society of Anesthesiology and Reanimation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: gemlikanesthesia
Record Dates: First submitted 2022-05-22; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Apnea; Hypoxia
Keywords: High Flow Nasal Oxygen; nasal cannula; colonoscopy
MeSH Terms: conditions — Apnea; Hypoxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard nasal therapy (Active Comparator): nasal oxygen was applied for procedure
  %40 inspired oxygen fraction five minutes preoxygenation
  Interventions: Device: High Flow Nasal Cannula
- high flow nasal cannula (Active Comparator): High Flow Nasal Oxygen was applied for procedure
  %40 inspired oxygen fraction five minutes preoxygenation
  Interventions: Device: High Flow Nasal Cannula

INTERVENTIONS:
Device: High Flow Nasal Cannula — high flow nasale cannula

SUMMARY:
Investigation of the Clinical Efficacy of High Flow Nasal Oxygen in Patients Over 60 Years of Age Undergoing Colonoscopy

DETAILED DESCRIPTION:
70 patients who underwent colonoscopy under elective conditions will be included in the study. Routine monitoring will be applied to the patients in the outpatient room in accordance with the standard protocol and the findings in the preoperative period will be recorded. The dose and frequency of anesthesia applied in the routine will not be interfered with and the recorded data will be collected by an observer other than the practitioner. Randomization between groups will be achieved by taking the patients on the surgical procedure list sequentially.

For both groups, after positioning the patients and placing the cannulas, preoxygenation will be performed for 5 minutes before induction of anesthesia. Oxygenation will be carried out at 35°C and 50 lt/min flow rate from the High Flow Nasal Cannula device, with inspired oxygen fraction equivalent to 40% in both groups, 5 lt/min in Group N, and inspired oxygen fraction equivalent to 40% in Group H, and immediately Anesthesia induction will then be applied.Oxygen saturation and other hemodynamic data of the patients in the room air before preoxygenation,oxygen saturation and hemodynamic data before induction after preoxygenation, oxygen saturation and hemodynamic data every minute during the procedure,oxygen saturation and hemodynamic data at the end of the procedure will be recorded. Interventions for respiratory safety, such as chin thrust, painful stimulus, inspired oxygen fraction increase, airway placement and mask ventilation, in case of apnea (stopping breathing for 10 seconds or more) or oxygen saturation ≤92% that may occur after induction until the end of the procedure , drug applications and other undesirable events will be recorded.

As a result of the study, High Flow Nasal Cannula and low flow nasal cannula, which is the standard conventional method, will be compared in terms of desaturation and hypoxemia in my colonoscopy procedures performed under sedation.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopy under elective conditions
* Patients aged 60 and over
* Having an American Society of Anesthesiology score of 1, 2, 3
* Approved and signed the informed consent form

Exclusion Criteria:

* Patients younger than 60 years
* Patients with an American Society of Anesthesiology score of 4 and above
* Emergency cases
* Patients who did not accept informed consent
* History of drug allergy and opioid tolerance
* Coagulation disorder
* Those who refused to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-26 (Estimated); Primary Completion 2022-11-12 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
hypoxia | during the procedure
  oxygen saturation <92
apnea | during the procedure
  spontaneous breathing not longer than 10 seconds

IPD SHARING:
Plan to Share IPD: Yes
researchers should explain the purpose of using individual participant data
Supporting Information: Study Protocol, CSR
Time Frame: when the study data is fully collected

REFERENCES:
- [Background] Riccio CA, Sarmiento S, Minhajuddin A, Nasir D, Fox AA. High-flow versus standard nasal cannula in morbidly obese patients during colonoscopy: A prospective, randomized clinical trial. J Clin Anesth. 2019 May;54:19-24. doi: 10.1016/j.jclinane.2018.10.026. Epub 2018 Nov 2. PMID 30391445
- [Background] Spence EA, Rajaleelan W, Wong J, Chung F, Wong DT. The Effectiveness of High-Flow Nasal Oxygen During the Intraoperative Period: A Systematic Review and Meta-analysis. Anesth Analg. 2020 Oct;131(4):1102-1110. doi: 10.1213/ANE.0000000000005073. PMID 32925331